CLINICAL TRIAL: NCT05966519
Title: ROSA Knee Intraoperative Planning Flexibility on Japan Preferred Surgical Technique, a Single Center Prospective Study
Brief Title: ROSA Knee Intraoperative Planning Flexibility Study
Acronym: IntraOP
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2022-29TDS
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Osteo Arthritis Knee; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- TKA with ROSA Knee: Total Knee Arthroplasty (TKA) is conducted using with robotic surgical assistant (ROSA) system
  Interventions: Device: Total Knee Replacement (TKR)

INTERVENTIONS:
Device: Total Knee Replacement (TKR) — Damaged cartilage of knee due to degenerative disease is replaced with metallic and plastic protheses

SUMMARY:
The purpose of this study is to verify that an orthopedic surgical assist robot (ROSA Knee System) can provide intraoperative adjustment of osteotomy angle and volume for total knee arthroplasty (TKA) based on feedbacks obtained from intraoperative soft tissue conditions. A total 80 cases will be enrolled at one study site with a postoperative follow-up period of 2 years.

DETAILED DESCRIPTION:
The objectives of the study are to document that ROSA Knee System can provide intraoperative planning adjustment based on feedbacks obtained by laxity as well as gaps to locally preferred surgeon's operative philosophy. This will also provide accuracy, intraoperative soft tissue release as well as patient outcome on locally preferred surgical technique.

The primary endpoint is defined as the mean absolute difference between X-Atlas image-based pre-op plan & intra-op final plan.

The secondary endpoints include Kinematic Analysis, EuroQol 5 dimensions (EQ-5D), Rehabilitation record, Knee Society Score (KSS) 2011, image assessment and Safety up to 2 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and over
* Skeletally matured
* Decision to have Total Knee Arthroplasty with ROSA Knee System being made independently and prior to recruitment into study
* Willing and able to complete scheduled follow-up evaluations as described in the study protocol
* Has participated in the informed consent process and is willing and able to sign an Institutional Review Board (IRB)/Ethics Committee (EC) approved informed consent form

Exclusion Criteria:

* Has serious bone defect(s), which require(s) metallic augment, synthetic bone or allograft
* Is septic, has an active infection or has osteomyelitis at the affected joint
* Has vascular insufficiency, muscular atrophy at the implant site or neuromuscular disease which might jeopardize the outcome of the surgery
* Has any concomitant disease which is likely to jeopardize the functioning or success of the implant
* Is known to be pregnant
* Is a prisoner, known alcohol or drug abuser or mentally incompetent or unable to understand what participation in this study entails
* Has a known sensitivity or allergy to one or more of the implanted materials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise of males and females who require primary total knee arthroplasty and satisfy the inclusion/exclusion criteria outlined in this section of the protocol. In order to avoid potential selection bias, each Investigator will offer study participation to each consecutive eligible patient presenting as a candidate for primary total knee arthroplasty using the commercially available Zimmer Biomet total knee systems. Eligible candidates who express interest in study participation will be offered Informed Consent.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The mean absolute difference between X-Atlas image based pre-op plan & intra-op final plan | Immediate post-operative
  The mean absolute difference between X-Atlas image-based pre-op plan and intra-op final plan in order to demonstrate the ability of the system to allow for intra-operative adjustments

SECONDARY OUTCOMES:
Pain, range of knee motion and functional performance | Preoperative, Postoperative 1.5 months (option), 3 months, 6 months, 12 months and 24 months
  The Knee Society Score 2011, and Physical Exam to evaluate pain, range of knee motion and functional performance
QOL | Preoperative, Postoperative 1.5 months (option), 3 months, 6 months, 12 months and 24 months
  Subject quality-of-life will be measured by the EuroQol 5 dimensions 5-level (EQ-5D-5L)
Rehabilitation record | Preoperative, Postoperative 1.5 months (option), 3 months, 6 months, 12 months and 24 months
  Recovery of patient will be assessed by prescribed Rehabilitation record and compliance
Kinematic analysis | Postoperative 12 months or 24 months
  Kinematic analysis will be conducted to visualize postoperative knee motion
Image review (CT/Radiograph) | Preoperative, Discharge, Postoperative 1.5 months (option), 3 months, 6 months, 12 months and 24 months
  Image review (CT/Radiograph) to assess the accuracy of the implant position, radiolucency, osteolysis, atrophy, hypertrophy, component migration, device fracture, heterotopic ossification, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yasuharu Nakashima, Principal Investigator — Kyushu University
Locations (1):
- Kyushu University Hospital, Fukuoka, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No